CLINICAL TRIAL: NCT05825365
Title: The Efficacy of Selumetinib in Chinese Paediatric Participants With Post-operative Neurofibromatosis Type 1 (NF1)-Associated PNs: A PhaseⅡ, Multicenter, Randomised, Double-Blinded, Placebo-Controlled Study
Brief Title: Selumetinib in Chinese Paediatric With Post-operative NF1-PNs, PhaseⅡ, Double-Blinded, Placebo-Controlled Study
Acronym: PROTECT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Selumetinib launch approval achieved in advance,strategy changesa new study will be generated in place of this study.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1346C00018
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Neurofibromatosis Type 1; Plexiform Neurofibromas; Post-operative
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — AZD 6244

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selumetinib (Active Comparator): Participants will orally receive selumetinib twice daily (BID) (approximately every 12 hours) at a dose of 25 mg per square meter of body surface area (BSA) on a continuous dosing schedule (28-day per cycle with no rest periods between cycles) for a maximum of 36 cycles.
  Interventions: Drug: Selumetinib
- Placebo (Placebo Comparator): Participants will orally receive placebo twice daily (BID) (approximately every12 hours) at a dose of 25 mg per square meter of body surface area (BSA) on a continuous dosing schedule (28-day per cycle with no rest periods between cycles) for a maximum of 36 cycles. Transfer to selumetinib on REiNS-defined PD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selumetinib — Selumetinib
  Arms: Selumetinib
Drug: Placebo — Placebo (Transfer to selumetinib on REiNS-defined PD)
  Arms: Placebo

SUMMARY:
This is a phase II, multicenter, randomised, parallel, double-blind, placebo-controlled study assessing the efficacy and safety of the MEKi selumetinib compared with placebo in Chinese paediatric participants with post-operative NF1-associated PNs.

DETAILED DESCRIPTION:
Participant Population:

The target population of interest in this study is Chinese paediatric participants with post-operative NF1-associated PNs who have received sub-total or partial resection of the targeted PN lesion (residue should be > 20% of pre-operative tumour volume, and measurable, defined as a lesion of ≥3 cm measured in one dimension on ≥3 imaging slices and have a reasonably well-defined contour), at least 4 weeks and up to 3 months after surgery.

Number of Participants:

Approximately 42 Chinese paediatric participants with post-operative NF1-associated PN will be randomised in a 2:1 ratio to receive selumetinib (28 participants) or placebo (14 participants).

Treatment Groups and Duration:

Following the screening period (Day -28 to Day -1), enrolled participants will be randomised in a 2:1 ratio to one of the treatment groups. Randomisation will be stratified by age (<12 versus ≥12 years old).

Participants will orally receive selumetinib or placebo twice daily (BID) (approximately every 12 hours) at a dose of 25 mg per square meter of body surface area (BSA) on a continuous dosing schedule (28-day per cycle with no rest periods between cycles) for a maximum of 36 cycles. Participants should be instructed to take the dose of selumetinib or placebo on an empty stomach (no food or drink other than water for 2 hours before and 1 hour after dosing) with water only. The capsules cannot be crushed and must be swallowed whole.

Dosing will be performed based on BSA calculated by the equation below, and doses will be rounded to the nearest 5 to 10 mg using a dosing nomogram. BSA should be calculated at screening and every tumour assessment visit. The dose of investigational medicinal product (IMP) will be capped at 50 mg when BSA is ≥1.9 m2.

All participants will be evaluated for safety and efficacy at a regular basis, as defined in Table 1. The safety follow-up visit will be conducted at Day 28 after the end of treatment (EOT) or treatment discontinuation.

Tumour assessments, measured by 3D volumetric magnetic resonance imaging will be determined by investigators according to REiNS criteria. Participants in the placebo group can be transferred to the selumetinib group within the study, when REiNS-defined progression of disease (PD) was detected in a participant. During the intervention period, participants may continue to receive selumetinib beyond REiNS-defined PD as long as they are continuing to show clinical benefit, as judged by the investigators and Sponsor.

Participants should continue on treatment until:

Unacceptable safety & tolerability event; Participants withdraw from the study; Completing 36 cycles of treatment or 24 cycles after last participant in (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

1. Paediatric subjects: Subjects ≥3 years and <18 years of age with a BSA ≥0.55 m2 at the time of study enrolment.
2. All study participants must have either positive genetic testing for NF1 or have at least one other diagnostic criterion for NF1 listed below Six or more macules (≥0.5cm in greatest diameter in pre-pubertal participants or ≥1.5 cm in greatest diameter in post-pubertal participants)； Freckling in the axillary or inguinal regions； Optic pathway glioma; Two or more iris Lisch nodules identified by slit lamp examination or 2 or more choroidal abnormalities-defined as bright, patchy nodules imaged by optical coherence tomography/near-infrared reflectance imaging; A distinctive bony lesion (such as: sphenoid dysplasia, anterolateral bowing of the tibia, or pseudoarthrosis of a long bone); A NF1 heterozygous pathogenic variant with a variant allele fraction of 50% in apparently normal tissue such as white blood cells; A parent with NF1 by the above criteria.
3. Symptomatic PNs:The PN has to cause or have the potential to cause significant clinical complications, as judged by the investigator, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, paraspinal lesions that can cause myelopathy brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) orare significantly disfiguring, lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions.

   A PN is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches. A spinal PN involves two or more levels with connection between the levels or extending laterally along the nerve.
4. All study participants have received sub-total or partial resection of the targeted PN lesion (residue should be > 20% of pre-operation volume, and measurable, defined as a lesion of ≥3 cm measured in one dimension on ≥3 imaging slices and have a reasonably well-defined contour), at least 4 weeks and up to 3 months after surgery.
5. Performance status: Subjects >16 years of age must have a Karnofsky performance level of ≥70, and children ≤16 years old must have a Lansky performance of ≥70 (Appendix G). Participants who are wheelchair bound or have limited mobility secondary to a need for mechanical breathing support (such as an airway PN requiring tracheostomy or continuous positive airway pressure) who must have a Lansky performance of ≥40 (Appendix G).
6. All participants must be able to swallow whole capsules.
7. Adequate organ and marrow function as follows with no blood transfusions (of red blood cells/ other blood products) within 28 days prior to screening assessment and no growth factors within 7 days prior to screening assessment:

   Haemoglobin ≥9.0 g/dL; Absolute neutrophil count ≥1.5×109/L; Platelet count ≥100×109/L; Total bilirubin (TBL) ≤1.5×the upper limit of normal (ULN) or ≤3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) - choose from below options: ALT and AST ≤2×ULN; Serum creatinine or calculated creatinine clearance - choose from below options: Serum creatinine >0.8 mg/dL for participants aged ≥1 to <4 years or >1.0 mg/dL for participants aged ≥4 years.
8. Reproduction:

   Negative pregnancy test (serum) for women of childbearing potential. Female participants must be 1 year post-menopausal, surgically sterile, or using one highly effective form of birth control (a highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly) Women of childbearing potential must agree to use one highly effective method of birth control. They should have been stable on their chosen method of birth control for a minimum of 3 months before entering the study and continue to use it throughout the study and until at least 7 days after the last dose.

   Non sterilised male partners of a woman of childbearing potential must use a male condom plus spermicide (condom alone in countries where spermicides are not approved) throughout this period and until at least one week after the female participant's last dose of study intervention. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant.

   Non-sterilised male participants (including males sterilised by a method other than bilateral orchidectomy e.g., vasectomy) who intend to be sexually active with a female partner of childbearing potential must be using an acceptable method of contraception such as male condom plus spermicide (condom alone in countries where spermicides are not approved) from the time of screening throughout the total duration of the study and the drug washout period (at least 7 days after the last dose of study intervention) to prevent pregnancy in a partner. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Vasectomised (i.e., sterile) males are considered fertile and should still use a male condom plus spermicide as indicated above during the clinical study. Even if the female partner is pregnant, male participants should still use a condom plus spermicide (where approved), as indicated above during the clinical study. Male participants must not donate or bank sperm during this same time period. Female partners (of childbearing potential) of male participants must also use a highly effective method of contraception throughout this period.
9. Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent. Parent/legal guardian consent is required in the assent process with appropriate documentation. Mandatory provision of signed and dated parent/legal guardian consent for the study along with the paediatric assent form, when applicable. For participants who reach the age of legal consent during the clinical study, notification may be required and a new consent form may need to be signed by the participant.

Exclusion Criteria:

1. Participants with confirmed or suspected malignant glioma or MPNST. Participants with low-grade gliomas (LGG) (including optic glioma) not requiring systemic therapy or radiation therapy are permitted.
2. History of malignancy except for malignancy treatment with curative intent with no known active disease ≥2 years before the first dose of study intervention and of low potential risk of recurrence.
3. Subjects with clinically significant cardiovascular disease as defined by the following:

   Known inherited coronary disease; Blood Pressure (BP): Uncontrolled hypertension (at screening: BP ≥140/90 mmHg despite optimal therapy); Acute coronary syndrome within 6 months prior to starting treatment; Uncontrolled angina - Canadian Cardiovascular Society grade II to IV despite medical therapy (Appendix F); Symptomatic heart failure New York Heart Association Class II to IV, prior or current cardiomyopathy, or severe valvular heart disease (Appendix F); Prior or current cardiomyopathy; Baseline left ventricular ejection fraction (LVEF) below the lower limit of normal (LLN) or <55% measured by echocardiogram or institution's LLN for multigated acquisition (MUGA); Severe valvular heart disease; Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication may be permitted upon discussion with the AstraZeneca Medical Monitor; QT interval corrected by Fridericia's method (QTcF) >470 ms or other factors that increase the risk of QT prolongation.
4. Subjects with the following ophthalmological findings/conditions:

   Current or past history of retinal pigment epithelial detachment/central serous retinopathy or retinal vein occlusion; Intraocular pressure >21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP). Subjects with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the Medical Monitor; Participants with any other significant abnormality on ophthalmic examination should be discussed with the Sponsor for potential eligibility.
5. Have received or are receiving an IMP or other systemic PN target treatment (including chemotherapy, immunotherapy, targeted therapy, biologic therapy or monoclonal antibodies) within 4 weeks prior to the first dose of study treatment, or within a period during which the IMP or systemic PN target treatment has not been cleared from the body (e.g. a period of 5 'half-lives'), whichever is longer.
6. Has received radiotherapy in the 6 weeks prior to the start of study intervention or any prior radiotherapy directed at the target or non-target PN.
7. Inability to undergo MRI and/or contraindication for MRI examinations. Prosthesis or orthopaedic or dental braces in close proximity to the area of interest that would interfere with volumetric analysis of target PN on MRI.
8. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of selumetinib.
9. Have had prior treatment with a MEK inhibitor.
10. Has received Vitamin E in the 7 days prior to initiation of IMP (does not apply to Granule formulation).
11. Receiving herbal supplements or medications known to be strong or moderate inhibitors or inducers of the cytochrome P450 (CYP)2C19 and CYP3A4 enzymes or fluconazole unless such products can be safely discontinued at least 14 days or 5 half-lives (whichever is longer) before the first dose of study medication.
12. Persistent toxicities (CTCAE Grade ≥2) caused by previous therapy for NF1-PN, excluding hair changes such as alopecia or hair lightening. If considered appropriate for a study then include: Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention may be included (e.g., hearing loss) after consultation with the AstraZeneca Medical Monitor.
13. Currently pregnant (confirmed with positive pregnancy test) or breastfeeding (lactation must be discontinued throughout the period of the study and until at least one week after the last dose of study intervention).
14. As judged by the investigator, any evidence of diseases such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant and active bleeding diseases which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardise compliance with the protocol.
15. Known severe hypersensitivity to selumetinib or any excipient of selumetinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib. For certain participant population, exceptions could also include carcinomas in situ or Ta tumours treated with curative intent.
16. Recent major surgery within a minimum of 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access.
17. Inability to swallow capsules, since capsules cannot be crushed or broken.
18. Clinical judgement by the investigator that the patient should not participate in the study.
19. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) Rate | 2 years
  The time from randomisation to MRI assessment of objective disease progression (PD) or death (by any cause in the absence of progression) per REiNS criteria. PD is defined as an increase in target PN volume by 20% or more compared to baseline or compared to the time of best response after documenting a partial response (PR). The appearance of new PN (with the exception of new discrete subcutaneous neurofibromas) or unequivocal progression of existing clinically relevant non-target PN is also considered PD.

SECONDARY OUTCOMES:
Confirmed Partial Response(cPR) Rate in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  Confirmed partial response (cPR) is the response of participants who have ≥20% decrease of target tumour volume from baseline confirmed by a consecutive scan within 3 to 6 months after the first response. Durable partial response (dPR) is cPR for at least 12 cycles of treatment. And CR is the response of participants who have the target lesion disappearance.
Durable Partial Response (dPR) rate in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  Durable Partial Response (dPR) rate is proportion of participants who have cPR for at least 12 cycles of selumetinib.
Complete Response (CR) rate in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  Complete Response (CR) rate is proportion of participants who have the target lesion disappearance.
Time to Initial Response in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  Time to Initial Response is the time between randomisation and the first PR.
Time to Best Response in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  Time to Best Response is the time between randomisation and the documented best efficacy evaluation (firstly occurs).
Tumour volume growth tracking | From begin to the end of treatment, around 2-3 years.
  A waterfall plot will present the largest percentages of decrease from baseline of tumour volume, as the tumour volumes growth tracking, with the auxiliary lines for -20% and 20%.
Health related quality of life (HRQoL) in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  In all participants who are randomised in the study, Health related quality of life (HRQoL) measured by Paediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales
Pain index in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  The FLACC scale is an observer-reported measurement used to assess pain in children aged from 2 months to 7 years, or for individuals that are unable to communicate their pain. In this study, parents will receive a short training on how to do the assessments of pain for their child.
Faces Pain Scale-Revised (4 to 17 years) in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  The Faces pain scale - revised is a self-reported measure of pain intensity developed for children. In this study, the Faces pain scale will be used to assess pain in children aged from 4 to 17 years of age.
Pain interference index in all participants who are randomised in the study. | From begin to the end of treatment, around 2-3 years.
  The Pain Interference Index (PII) is a six-item measure that assesses the degree to which pain has interfered with daily activities in the past week, including paying attention, spending time with friends, doing leisure and physical activities, mood, and sleep. In this study, the Faces pain scale will be used to assess pain in children aged from 4 to 17 years of age. If participants have difficulties reading, it is permissible for site staff to read the instructions to the participant and point to the faces as they read the instructions. If a participant has difficulties remembering the worst pain they had the past week, instructions should be given to assess the worst pain they had today.
Pain Medication Survey (All Participants) | From begin to the end of treatment, around 2-3 years.
  A pain medication survey will be used to ensure that potential pain palliation is not the result of increased usage of analgesics.Information on daily and as-needed pain medications will be collected, including dates, pain medication name, dose and frequency.
Strength and Range of Motion | From begin to the end of treatment, around 2-3 years.
  Manual muscle testing was performed by a physiatrist or physical therapist to determine the strength of specific muscle groups at each restaging visit using the Medical Research Council 0-5 strength scale.
Disfigurement in all Consenting participants. | From begin to the end of treatment, around 2-3 years.
  Consenting participants will have photographic documentation of visible PNs.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ni, Principal Investigator — Beijing Children's Hospital